CLINICAL TRIAL: NCT01274637
Title: Postpartum Prophylaxis for PE Randomized Control Trial Pilot: A Pilot Study Assessing Feasibility of a Randomized, Open-label Trial of Low-Molecular-Weight-Heparin for Postpartum Prophylaxis in Women at Risk of Developing Venous Thromboembolism
Brief Title: PROSPER: PostpaRtum PrOphylaxiS for PE Randomized Control Trial Pilot
Acronym: PROSPER
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ottawa Hospital Research Institute (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2010303-01H
Record Dates: First submitted 2011-01-10; First posted 2011-01-11 (Estimated); Results first posted 2017-08-01 (Actual); Last update posted 2017-08-01 (Actual); Status verified 2017-01

CONDITIONS: Venous Thromboembolism; Postpartum
Keywords: postpartum; low molecular weight heparin; venous thromboembolism; prophylaxis; Dalteparin Sodium
MeSH Terms: conditions — Venous Thromboembolism | interventions — Dalteparin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- low molecular weight heparin (Experimental): Prophylactic-dose (5000 IU/0.2ml)low molecular weight heparin (LMWH), administered subcutaneously once daily in pre-filled glass syringes for 10 days (+/- 3 days) for a total of 10 (+/-3) study drug injections.
  Interventions: Drug: Dalteparin Sodium
- Control Group (No Intervention): No treatment control group.

INTERVENTIONS:
Drug: Dalteparin Sodium — 5,000 IU/0.2ml (anti-Xa) administered once daily in prefilled glass syringes.
  Other Names: Fragmin; Dalteparin Sodium(DIN 02132648/NDC# 62856-500)
  Arms: low molecular weight heparin

SUMMARY:
The purpose of this study is to determine if it is feasible to conduct a multi-center randomized trial to determine whether a blood thinner, low-molecular-weight-heparin (LMWH), is effective at preventing blood clots, thromboembolism (VTE), in postpartum women at risk.

DETAILED DESCRIPTION:
The PROPSER pilot is a randomized, open-label pilot study comparing prophylactic low molecular weight heparin (LMWH) to saline placebo. The PROSPER pilot study will assess the feasibility of conducting a full trial as measured by the number of subjects recruited per center per month. In addition, clinical data will be collected to determine an estimate of the primary outcome event rate (symptomatic VTE or asymptomatic proximal deep vein thrombosis (DVT) and major bleeding event rate for the full trial in LMWH and control groups. If our pilot results indicate that no substantial changes are needed to the study design, we will include the pilot data in the primary and secondary outcome analyses for the full trial (i.e. a "Vanguard trial" or internal pilot trial).

Eligible consenting women at risk of postpartum thrombosis will be randomized within 36 hours after delivery of the placenta and will be equally allocated to 2 trial arms, either the treatment group: prophylactic-dose LMWH, subcutaneously once daily for 10 days (+/-3 days), or the control group.

At 10 days (+/- 3 days), all women will have a study visit to assess for study outcomes, including bilateral leg ultrasound screening for VTE and a D-dimer test. A final telephone follow-up will occur at 90 days for outcome assessment of subsequent VTE, bleeding or other adverse events.

ELIGIBILITY:
Inclusion Criteria:

Women must be at high risk for thromboembolism for one of the following reasons:

1. Known low risk thrombophilia (Known = diagnosed prior to enrollment and low risk thrombophilia includes heterozygous factor V Leiden or prothrombin gene variant or protein C deficiency or protein S deficiency. If not previously tested then assumed not to have thrombophilia).
2. Immobilization (defined as >90% of waking hours in bed, of a week or more at any point in the antepartum period).

OR any two of the following reasons:

1. Postpartum infection (fever (temperature>38.5oC) and clinical signs/symptoms of infection and elevated neutrophil count (higher than local lab normal))
2. Postpartum hemorrhage (Estimated blood loss >1000 ml during delivery and postpartum)
3. Pre-pregnancy BMI >25 kg/m2
4. Emergency cesarean birth (emergency = not planned prior to onset of labour)
5. Smoking >5 cigarettes per day prior to pregnancy
6. Preeclampsia (blood pressure ≥ 140mmHG systolic and/or ≥90 mmHg diastolic on at least one occasion and proteinuria (1+ on urine dipstick or 300mg/dl or total excretion of 300mg/24 hours) or typical end-organ dysfunction.
7. Infant birth weight (adjusted for sex and gestational age) <3rd percentile (i.e., small for gestational age).

Exclusion Criteria:

1. Less than 6 hours or more than 36 hours since delivery at the time of randomization
2. Need for anticoagulation as judged by the local investigator, may include but not limited to:

   1. Personal history of previous provoked or unprovoked VTE (DVT or PE)
   2. Continuation of LMWH that was started in the antenatal period for VTE prophylaxis
   3. Mechanical heart valve
   4. Known high-risk thrombophilia (Known = diagnosed prior to enrolment and high-risk thrombophilia includes deficiency of antithrombin (at least 1 abnormal lab result), persistently positive anticardiolipin antibodies (> 30U/ml on two measurements a minimum of six weeks apart), persistently positive Anti B2 glycoprotein antibodies (> 20U/ml on two measurements a minimum of six weeks apart), persistently positive lupus anticoagulant (positive on two measurements a minimum of six weeks apart), homozygous factor V Leiden (FVL), homozygous prothrombin gene mutation (PGM), compound heterozygosity factor V Leiden (FVL) and prothrombin gene mutations (PGM), more than 1 thrombophilia (any combination of 2 or more: FVL, PGM, protein C deficiency, protein S deficiency). If not previously tested then assumed not to have thrombophilia).
3. Contraindication to heparin therapy, including:

   1. History of heparin induced thrombocytopenia (HIT)
   2. Platelet count of less than 80,000 x 106/L on postpartum Complete Blood Count(CBC)
   3. Hemoglobin ≤ 75 g/L on postpartum CBC
   4. Active bleeding at any site (not resolved prior to randomization)
   5. Excessive postpartum vaginal bleeding (>1 pad per hour prior to randomization).
   6. Documented gastrointestinal ulcer within 6 weeks prior to randomization
   7. History of heparin or LMWH allergy
   8. Severe postpartum hypertension (systolic blood pressure (SBP) > 200mm/hg and/or diastolic blood pressure (DBP) > 120mm/hg)
   9. Severe hepatic failure (INR >1.8 if liver disease suspected)
4. Have received more than one dose of heparin or LMWH since delivery
5. < age of legal majority in local jurisdiction (age <18 in Canada)
6. Prior participation in PROSPER
7. Unable or refused to consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2011-03; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc A Rodger, M.D., MSc., Principal Investigator — Ottawa Hospital Research Institute
Locations (7):
- United States (2):
  - University of Virginia Medical Center, Charlottesville, Virginia
  - Puget Sound Blood Center, Seattle, Washington
- Canada (5):
  - Royal Alexandra Hospital, Edmonton, Alberta
  - McMaster University Medical Centre, Hamilton, Ontario
  - Ottawa Hospital General Campus & Civic Campus, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - SMBD Jewish General Hospital, Montreal, Quebec

REFERENCES:
- [Result] Rodger MA, Phillips P, Kahn SR, Bates S, McDonald S, Khurana R, James AH, Konkle BA; PROSPER Investigators: Tim Ramsay, Dean Fergusson, Anne McLeod, Wee Shian Chan, Rshmi Khurana, Kara Narenberg, Haim Abenhaim, John Heit, Ghada Bourjeilly, Paul Gibson, Kent Bailey. Low molecular weight heparin to prevent postpartum venous thromboembolism: A pilot study to assess the feasibility of a randomized, open-label trial. Thromb Res. 2016 Jun;142:17-20. doi: 10.1016/j.thromres.2016.04.004. Epub 2016 Apr 9. No abstract available. PMID 27096813
- [Result] Rodger MA, Phillips P, Kahn SR, James AH, Konkle BA; PROSPER Investigators. Low-molecular-weight heparin to prevent postpartum venous thromboembolism. A pilot randomised placebo-controlled trial. Thromb Haemost. 2015 Jan;113(1):212-6. doi: 10.1160/TH14-06-0485. Epub 2014 Nov 6. PMID 25373438
- [Derived] Middleton P, Shepherd E, Gomersall JC. Venous thromboembolism prophylaxis for women at risk during pregnancy and the early postnatal period. Cochrane Database Syst Rev. 2021 Mar 29;3(3):CD001689. doi: 10.1002/14651858.CD001689.pub4. PMID 33779986

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Potential subjects were initially approached by a member of the health care team providing their care (physician, nurse, care facilitator, etc.). If the patient agreed to being contacted, the Investigator or designate provided detailed information regarding the study and assessed the individual's eligibility for the study.
Period: Overall Study
Arm/Group | Low Molecular Weight Heparin | Control Group
Started | 30 | 32
Completed | 30 | 30
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Molecular Weight Heparin | Control Group | Total
Number analyzed (Participants) | 30 | 32 | 62
Age, Continuous [Mean (Full Range); unit: years] | 30.0 [20 to 43] | 31.6 [18 to 38] | 30.8 [18 to 43]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 32 | 62
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 28 | 30 | 58
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 2 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 3 | 7
  White | 24 | 27 | 51
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Canada | 27 | 28 | 55
  United States | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of Recruitment and Trial Operations.
Description: The average number of subjects that are recruited per site per month during a 4 month active recruitment phase at each site.
Time Frame: 4 months
Measure: Number; unit: participants per site per month
Arm/Group | Low Molecular Weight Heparin | Control Group
Number analyzed (Participants) | 30 | 32
participants per site per month | 0.9 | 0.9

2. Secondary Outcome: Venous Thromboembolism in the Early Postpartum Period.
Description: This includes symptomatic Deep Vein Thrombosis (DVT) or pulmonary embolism (PE) in the interval between randomization and the last dose of study drug (10 days +/- 3 days) OR asymptomatic proximal DVT detected by compression ultrasound of both legs done within 24hrs of the last dose of study drug (10 days (+/- 3 days) postpartum). Compressed and non-compressed images will be obtained from the calf trifurcation to the inguinal ligament. All suspected outcomes will be adjudicated by a blinded expert adjudication committee.
Time Frame: From randomization to Day 10
Measure: Count of Participants; unit: Participants
Arm/Group | Low Molecular Weight Heparin | Control Group
Number analyzed (Participants) | 30 | 30
Participants | 0 | 0

3. Secondary Outcome: Late Symptomatic Venous Thromboembolism
Description: This includes symptomatic Deep Vein Thrombosis or Pulmonary Embolism. Suspected outcomes will be adjudicated by a blinded adjudication committee.
Time Frame: From Day 10 to Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | Low Molecular Weight Heparin | Control Group
Number analyzed (Participants) | 30 | 30
Participants | 0 | 0

4. Secondary Outcome: Death From Venous Thromboembolism
Description: If a subject dies between randomization and late postpartum follow up (Day 90 +/- 7 days) the death will be adjudicated as certain, highly probable, probable, or unlikely due to Pulmonary Embolism (PE) using the following criteria.
  Certain: hypotension, hypoxia, cardiac arrest with no other explanation other than PE and autopsy or radiographic confirmation Highly probable: criteria for certain but another disease could have caused the death Probable: other cause suspected based on clinical evidence but 100% certainty not available Unlikely: all other cases.
Time Frame: From Randomization to Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | Low Molecular Weight Heparin | Control Group
Number analyzed (Participants) | 30 | 32
Participants | 0 | 0

5. Secondary Outcome: Major Bleeding or Clinically Relevant Non-major Bleeding
Description: Major bleeding meets at least one of the following: Fatal bleeding; Symptomatic bleeding in a critical area or organ (intracranial, intraspinal, retroperitoneal, etc.); Bleeding causing a fall in hemoglobin level of 20 g L-1 (1.24 mmol L-1) or more, or leading to transfusion of two or more units of whole blood or red cells .
  Clinically Relevant Non-major Bleeding does not meet the criteria for major bleeding but meets at least one of the following: Hospitalization; Medical intervention; Unscheduled contact with a physician; Discomfort (pain, or impairment of activities of daily life).
Time Frame: From Randomization to Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | Low Molecular Weight Heparin | Control Group
Number analyzed (Participants) | 30 | 32
Participants | 3 | 1

6. Secondary Outcome: Heparin Induced Thrombocytopenia
Description: All subjects who develop thrombocytopenia (platelets less than 80 x 109/L and/or with >50% decrease from baseline) will be investigated for Heparin Induced Thrombocytopenia (HIT) by having ELISA and serotonin release assays to confirm or refute a diagnosis of HIT. HIT will be diagnosed with a positive PF4 (platelet factor 4) HIT ELISA assay.
Time Frame: From Randomization to Day 90
Measure: Count of Participants; unit: Participants
Arm/Group | Low Molecular Weight Heparin | Control Group
Number analyzed (Participants) | 30 | 32
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Low Molecular Weight Heparin | Control Group
Serious Adverse Events (participants affected / at risk) | 2/30 | 0/32
Other Adverse Events (participants affected / at risk) | 3/30 | 0/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Molecular Weight Heparin (N=30) | Control Group (N=32)
Hospitalization (Pregnancy, puerperium and perinatal conditions) | 1 | 0 — Hospitalization for post-partum bleeding event
Hospitalization (Infections and infestations) | 1 | 0 — Hospitalization for post-partum infection
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Molecular Weight Heparin (N=30) | Control Group (N=32)
Cellulitis (Infections and infestations) | 1 | 0 — Cellulitis of c-section incision
Cellulitis (Infections and infestations) | 1 | 0 — Cellulitis of left lower leg, resolving with antibiotics
Abnormal Lab result (Blood and lymphatic system disorders) | 1 | 0 — Critically low hemoglobin

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No